CLINICAL TRIAL: NCT03467607
Title: A Feasibility Study of a Low Tidal Volume Ventilation Strategy in One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, ignacio martin loeches, Consultant Intensivist, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-11 List 43 (1)
Record Dates: First submitted 2018-01-19; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Low Tidal Volume Ventilation

STUDY DESIGN:
Intervention Model Description: parallel assignment
Masking Description: open label, randomisation blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3ml/kg (Active Comparator): 15 patients ventilated with 3ml/kg ideal body weight while on one lung ventilation
  Interventions: Procedure: tidal volume ventilation
- 4ml/kg (Active Comparator): 15 patients ventilated with 4ml/kg ideal body weight while on one lung ventilation
  Interventions: Procedure: tidal volume ventilation
- control (Active Comparator): 15 patients ventilated using the anaesthetists usual ventilation strategy
  Interventions: Procedure: tidal volume ventilation

INTERVENTIONS:
Procedure: tidal volume ventilation — low tidal volume ventilation

SUMMARY:
A study of two ventilatory strategies for low tidal volume ventilation compared to a control group to elucidate if low tidal volumes of 3ml/kg or 4ml/kg were feasible for one lung ventilation.

DETAILED DESCRIPTION:
This study investigated the feasibility of low tidal volume ventilation for one lung ventilation.

45 patients were recruited - 15 patients in each of three groups, 3ml/kg, 4ml/kg or usual care.

Outcomes studied were length of stay, 30 day mortality, unplanned ICU admission, evidence of respiratory failure or requirement for non-invasive ventilation, chest x-ray infiltrates and requirement for antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III lung resection surgery requiring one lung ventilation

Exclusion Criteria:

* ASA IV or above under 18 or over 80 years of age pregnancy previous lung lobectomy or pneumonectomy requirement for massive transfusion during the case BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Radiological evidence of injury to the ventilated lung | post operatively up to 6 weeks post operatively
  evidence of infiltrates in the non operative lung
unplanned ICU admission | up to 6 weeks post operatively
  unplanned admission to the icu with respiratory issues
Requirement for non-invasive ventilation | up to 6 weeks post operatively
  whether a patient in the trial requires niv for respiratory failure
Hospital acquired pneumonia | up to discharge at 6 weeks post operatively
  pneumonia acquired in hospital

SECONDARY OUTCOMES:
length of hospital stay | until patient discharge at 6 weeks post operatively
  number of days in hospital
length of icu stay | until patient discharge at 6 weeks post operatively
  number of days in ICU
30 day mortality | 30 days post operatively
  number of patients who died within 30 days of their procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Martin-Loeches, md, Study Chair — University of Dublin, Trinity College
Locations (1):
- St James's Hospital Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No